CLINICAL TRIAL: NCT01580683
Title: Effect of Ascorbic Acid on the Incidence of Post-operative Atrial Fibrillation in Patients Undergoing Cardiac Surgery
Brief Title: Vitamin C and Atrial Fibrillation After Cardiac Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No funding obtained to support patient recruitment
Sponsor: Regional Hospital of Scranton (Other)
Responsible Party: Principal Investigator, Scott Bolesta, Pharm.D., BCPS, Associate Professor or Pharmacy Practice and Clinical Pharmacist, Internal Medicine/Critical Care, Regional Hospital of Scranton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WU0811SB
Record Dates: First submitted 2012-04-13; First posted 2012-04-19 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Ascorbic Acid; Thoracic Surgery; Cardiac Arrhythmias; Cardiac Surgery; Vitamin C; Postoperative Complications; Antioxidants; Inflammation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Postoperative Complications; Inflammation | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ascorbic acid (Experimental)
  Interventions: Drug: Ascorbic Acid
- Placebo (Placebo Comparator)
  Interventions: Other: Identical Placebo

INTERVENTIONS:
Drug: Ascorbic Acid — Two 1 g capsules the evening prior to surgery, followed by one 1 g capsule every 12 hours starting the morning of the first postoperative day for 5 days.
  Other Names: Vitamin C
  Arms: Ascorbic acid
Other: Identical Placebo — Two capsules the evening prior to surgery, followed by one capsule every 12 hours starting the morning of the first postoperative day for 5 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if vitamin C decreases the chance of developing atrial fibrillation, a type of arrhythmia or irregular heartbeat, following cardiac surgery. This irregular heartbeat is a common occurrence following cardiac surgery, and occurs in about one third of patients. It poses extra risks to people who develop it. Our hypothesis is that Vitamin C will decrease the incidence of postoperative atrial fibrillation.

DETAILED DESCRIPTION:
The development of atrial fibrillation (AF) following cardiac surgery is relatively common, occurring in approximately 25-60% of patients. Coronary artery bypass graft surgery (CABG) carries the lowest risk of AF development, with an incidence of approximately 25-30%, followed by cardiac valve and combined CABG/cardiac valve surgeries, with incidences up to 60%. AF development in patients undergoing cardiac procedures has been linked to increases in postoperative morbidity and mortality, including an increase in readmission to the ICU, stroke, reintubation, and 30-day and 6-month mortality. Patients who develop AF have also been shown to experience longer hospital stays, both in the ICU and overall.

While some other medications have been shown to decrease the risk of AF development, the use of beta-blockers peri- and postoperatively have shown the most promise, and are the standard of care for patients undergoing CABG surgery. However, patients experiencing AF have been shown to experience cardiac production of peroxynitrite, corresponding to a hypothesis that AF occurs through oxidative stress. Due to this correlation, supplementation of ascorbate has been proposed as a treatment to reduce the risk of AF development following cardiac surgery. Ascorbate is a potent peroxynitrite antagonist, and may therefore reduce oxidative stress and AF development following cardiac surgery. This trial aims to assess the efficacy of ascorbic acid in reducing the incidence of postoperative AF in patients undergoing elective or urgent CABG surgery, cardiac valve surgery, or a combination of the two. Our hypothesis is that ascorbic acid will decrease the incidence of postoperative AF development.

ELIGIBILITY:
Inclusion Criteria:

* Adults 50 years of age or older
* Undergoing elective or urgent coronary artery bypass graft surgery, valve surgery, or a combination of the two

Exclusion Criteria:

* Prior cardiac surgery
* History of atrial fibrillation
* Permanent or temporary pace maker
* Currently taking digoxin or Vaughan Williams Class I or III antiarrhythmic medications
* Known hyperoxaluria
* History of renal calculi
* History of allergic or hypersensitivity reaction to ascorbic acid products
* Currently taking 1 g or more of ascorbic acid supplementation daily

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Post-operative atrial fibrillation | Patients will be followed for the entire hospital stay, with an expected average of 5 days

SECONDARY OUTCOMES:
Hospital length of stay | 30 Days
Intensive care unit length of stay | 30 Days
Stroke | 30 Days
Transient ischemic attack | 30 Days
Mortality | 30 Days
Hospital Readmission for atrial fibrillation | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Scott Bolesta, Pharm.D., Principal Investigator — Wilkes University
Locations (1):
- Regional Hospital of Scranton, Scranton, Pennsylvania, United States